CLINICAL TRIAL: NCT06370520
Title: Screening Emotions in Adolescents Receiving Care at the Hospital for mTBI (SEARCH-mTBI)
Brief Title: Screening Emotions in Adolescents at the Hospital for mTBI
Acronym: SEARCH-mTBI
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Pediatric Emergency Care Applied Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: 2122025
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Brain Injury Traumatic Mild; Brain Injuries; Brain Injuries, Acute; Head Injury With Intracranial Hemorrhage; Head Injury Trauma; Brain Injury Traumatic Focal With Loss of Consciousness; Skull Fractures; Diffuse Axonal Injury; Intracranial Hemorrhages; Head Injury
Keywords: Child; Concussion; Wounds and Injuries; Brain Injuries; Head Injuries Trauma; Loss of Consciousness
MeSH Terms: conditions — Brain Concussion; Brain Injuries; Intracranial Hemorrhage, Traumatic; Skull Fractures; Diffuse Axonal Injury; Intracranial Hemorrhages; Craniocerebral Trauma; Wounds and Injuries; Unconsciousness | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation Cohort: Four sites will enroll a derivation cohort (n=1512) of head-injured children. Qualified participants will complete or be evaluated with validated questionnaires. Data related to the mTBI event and the participants medical history will be recorded.
  Interventions: Behavioral: Validated Questionnaires; Behavioral: Questionnaires; Other: Clinician / Medical Record Variables
- Validation Cohort: Three sites will enroll a validation cohort (n=1080) of head-injured children. Qualified participants will complete or be evaluated with validated questionnaires. Data related to the mTBI event and the participants medical history will be recorded.
  Interventions: Behavioral: Validated Questionnaires; Behavioral: Questionnaires; Other: Clinician / Medical Record Variables

INTERVENTIONS:
Behavioral: Validated Questionnaires — Generalized Anxiety Disorder-7 (GAD-7), Patient Health Questionnaire-8 (PHQ-8), The Rivermead Post Concussion Symptom Questionnaire (Rivermead), Pediatric Quality of Life Inventory (PedsQL), Strengths and Difficulties Questionnaire (SDQ)
Behavioral: Questionnaires — Early Physical Activity/Return to School Questionnaire, Mental Health Utilization Questionnaire
Other: Clinician / Medical Record Variables — Medical History, Emergency Department Clinical Variables

SUMMARY:
The goal of this observational study is to develop and validate a clinical tool to predict which adolescents aged 11 to less than 18 years of age with mild traumatic brain injury (mTBI) are at an increased risk for developing significant new or worsening mental health conditions.

The main aims the study wish to answer are:

* Does the adolescent have new or worsening depression or anxiety defined as a change from their previous medical history using self-reported questionnaires at either one or three months post-injury?
* Does the adolescent have unmet mental health care needs, defined as not receiving any mental or behavior health care in patients with new or worsening anxiety or depression as defined by the self reported questionnaires?

Participants will be enrolled after being diagnosed in the emergency department (ED) with an mTBI. During the ED visit, the child's parent/caregiver and the adolescent will complete several questionnaires related to mental health which include tools to measure anxiety and depression. Participants will be asked to complete these questionnaires again at 1 month and 3 months post enrollment.

DETAILED DESCRIPTION:
This is an observational, multicenter study to develop and validate a clinical tool to predict mental health problems in adolescents (after mild traumatic brain injuries (mTBI).

The primary objective of the study is to develop and validate a clinical tool to predict which adolescents with mTBIs are at an increased risk for developing significant new or worsening mental health conditions. The investigators believe that at completion of this study they will have developed and validated a clinical prediction tool that will help clinicians define adolescents with mTBIs by risk of follow up mental health complications into low, moderate, and high-risk categories. This will provide clinicians with distinct risk categories on which make decisions about an adolescents care.

The investigators will also evaluate racial, ethnic, and social and economic differences in post-mTBI management across diverse populations of adolescents with mTBIs. The investigators believe that specific racial, ethnic, social, and economical characteristics will also be associated with unmet mental health needs in adolescents with mTBIs.

ELIGIBILITY:
Inclusion Criteria:

Children 11 to less than 18 years old who meet the Centers for Disease Control and Prevention (CDC) definition of mTBI*. In brief, this is defined as a Glasgow Coma Scale (GCS) score of 13 to 15 with:

- Head injury (e.g., direct blow or sudden deceleration/acceleration) plus any neurological sign and/or symptom such as headache, nausea, history of loss of consciousness, confusion, dizziness, amnesia (not limited to these symptoms/signs)

AND/OR

- Traumatic intracranial abnormalities on CT or MRI (such as intracranial hemorrhage, skull fracture, or diffuse axonal injury)

*mTBI is defined as an acute brain injury resulting in neurological symptoms such as confusion or disorientation, headache, nausea, loss of consciousness, amnesia, seizure, focal signs or symptoms, and/or have traumatic intracranial abnormalities on CT or MRI imaging. mTBI patients have GCS scores of 13 to 15. Per CDC precedent, we will use the term mTBI which encompasses other commonly used terms such as "concussion" or "minor head injury". This will include patients who may have neuroimaging findings of traumatic abnormalities (e.g., intracranial hemorrhage, diffuse axonal injury, skull fractures) which are risk factors for mental health problems; however, neuroimaging is not required for enrollment into the study.

Exclusion Criteria:

* Presentation to the ED >72 hours post-injury
* TBI requiring emergent neurosurgical intervention at the time of enrollment
* Other injuries requiring emergent surgery at the time of enrollment
* Parent or child unable to accurately complete the study questionnaires due to preexisting functional limitations (e.g., severe developmental delay)
* Previous known enrollment into the study
* Patient or parent does not speak English or Spanish

Ages: 11 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Participants are injured children aged 11 to 17 years old who present with a Mild traumatic brain injury (mTBI), including concussion, as defined by the Centers for Disease Control and Prevention as an acute brain injury resulting in neurological symptoms such as confusion or disorientation, loss of consciousness, amnesia, seizure, or other signs or symptoms combined with a Glasgow Coma Scale (GCS) score of 13 to 15 to one of six emergency departments (EDs) throughout the United States.
Sampling Method: Non-Probability Sample
Enrollment: 2592 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
New or worsening depression or anxiety | The Generalized Anxiety Disorder-7 (GAD-7) and Patient Health Questionnaire-8 (PHQ-8) are measured at approximately 30 days and approximately 90 days after the emergency department (ED) baseline visit.
  New or worsening depression or anxiety are binary variables (yes/no) defined as a change from the retrospective baseline score collected on the self-reported Generalized Anxiety Disorder-7 questionnaire (GAD-7) equal to or greater than 4 points, and/or a change from the baseline score collected on the self-reported Patient Health Questionnaire-8 (PHQ-8) equal to or greater than 5 points.
  The Generalized Anxiety Disorder-7 (GAD-7) contains seven items, each of which is scored 0 to 3, providing a 0 to 21 severity score where higher values indicate worsening severity.
  The Patient Health Questionnaire-8 (PHQ-8) contains eight items, each of which is scored 0 to 3, providing a 0 to 24 severity score where higher values indicate worsening severity.
Unmet mental health care needs in patients with new or worsening depression or anxiety | The Mental Health Utilization Questionnaire is completed at approximately 30 days and approximately 90 days after the emergency department (ED) baseline visit.
  Unmet mental health care needs are defined as a binary variable (yes/no) if participants received any mental or behavioral health care as collected on the self-reported Mental Health Utilization Questionnaire completed the parent of the participant. Mental or behavioral health care includes, but is not limited to behavioral, cognitive-behavioral, interpersonal therapy, psychotherapy, and counseling. Medications alone will not fulfill the criteria of mental or behavior health care.

SECONDARY OUTCOMES:
Decline in quality of life | The Pediatric Quality of Life Inventory Questionnaire (PedsQL) is measured at approximately 30 days and approximately 90 days after the emergency department (ED) baseline visit.
  A decline in the patient's quality of life is a binary variable (yes/no) defined as a decrease from the retrospective baseline score collected on the self-reported Pediatric Quality of Life Inventory questionnaire (PedsQL) equal to or greater than a 4.5 points.
  The Pediatric Quality of Life Inventory questionnaire (PedsQL) contains 23 items, each of which is scored 0 to 4, and is scored on a range from 0 to 100, with lower scores indicated a lower quality of life.
Persistent mTBI symptoms | The Rivermead Post Concussion Questionnaire is measured at approximately 30 days and approximately 90 days after the emergency department (ED) baseline visit.
  Persistent mTBI is a binary variable (yes/no) defined as an increase from the retrospective baseline score collected on the Rivermead Post Concussion Questionnaire of greater than or equal to 2 points on any three symptoms.
  The Rivermead Post Concussion Questionnaire consists of the sixteen items divided into two groups. The first three items make up the first sub-group scored from 0 to 12, and the next 13 items make up the second sub-group scored from 0 to 52. The entire questionnaire is scored from 0 to 64 where higher values indicate worsening severity.
New deficits in emotional/behavioral functioning or hyperactivity/inattention | The Strengths and Difficulties Questionnaire (SDQ) is measured at approximately 30 days and approximately 90 days after the emergency department (ED) baseline visit.
  The Strengths and Difficulties Questionnaire (SDQ) is comprised of 4 sub scales of 5 items each for a total of 20 questions. Each sub scale has a minimum score of 0 and a maximum score of 10 where higher values indicate worsening severity.
  New deficits in emotional/behavioral functioning or participant hyperactivity/inattention are binary variables (yes/no) defined as a new score of 5 points or greater on the emotional/behavioral functioning sub scales or 6 points or greater on the hyperactivity/inattention sub scale as collected from the self-reported Strengths and Difficulties Questionnaire (SDQ).
Parent Perception of Unmet Mental Health Needs | The Mental Health Utilization Questionnaire is completed at approximately 30 days and approximately 90 days after the emergency department (ED) baseline visit.
  Parent Perception of Unmet Mental Health Needs is a binary variable (yes/no) defined as the parent perception of unmet mental health needs in participants with new or worsening anxiety or depression identified at the 1 month and 3 month follow up visits. This will be assessed using the Mental Health Utilization Questionnaire completed by parents.
  Unmet mental health care needs are defined as a binary variable (yes/no) if participants received any mental or behavioral health care as collected on the self-reported Mental Health Utilization Questionnaire completed the parent of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K Nishijima, MD, MAS, Principal Investigator — University of California, Davis
Locations (6):
- United States (6):
  - University of California, Davis Medical Center, Sacramento, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hasbro Children's Hospital and Brown University, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Texas Children's Hospital, Houston, Texas
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No